CLINICAL TRIAL: NCT07384351
Title: Added Value of MRI Volumetry and Diffusion Tensor Imaging Over Conventional MRI in Temporal Lobe Epilepsy
Brief Title: MRI Volumetry and Diffusion Tensor Imaging in Temporal Lobe Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Saad EL Shazly, DR, Assiut University
Other Study IDs: MRI Volumetry, DTI in epilepsy
Record Dates: First submitted 2026-01-12; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Temporal Lobe Epilepsy (TLE)
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — MRI volumetry and Diffusion Tensor Imaging

SUMMARY:
This works aims at evaluating the diagnostic performance of combined MRI Volumetry, Diffusion tensor imaging and Conventional MRI in lateralizing the epileptogenic focus in patients with temporal lobe epilepsy and correlate these findings with clinical outcome.

DETAILED DESCRIPTION:
Epilepsy is one of the most common neurological diseases. It affects about 70 million people worldwide. Temporal lobe epilepsy (TLE) is the most common focal epilepsy and its most frequent cause is hippocampal sclerosis. Approximately one-third of patients with TLE have seizures which fail to respond to drug therapy and they require surgical resection of the epileptic focus. Drug resistant epilepsy (DRE) is associated with neurocognitive and psychological decline, poor quality of life, increased risk of premature death and higher economic burden.

Diagnosis of TLE typically relies on clinical evaluation, MRI to visualize affected areas, such as hippocampal sclerosis and EEG to detect abnormal electrical activity in the temporal lobe's cortical regions. However, both EEG and conventional MRI have limitations. About thirty percent of temporal lobe epilepsy (TLE) cases are negative on MRI, so quantitative diagnosis based on clinical symptoms becomes challenging.

The development of automatic MR volumetry makes it possible to account for hippocampal volume differences that may escape visual detection. MRI volumetry enables to objectively quantify brain volume changes associated with neurological conditions such as Alzheimer's disease, multiple sclerosis and epilepsy. Automated segmentation tools facilitate precise and reproducible analysis of structural brain changes, contributing significantly to early diagnosis, patient monitoring, and therapeutic planning. Progress in neuroimaging has led not only to successful identiﬁcation of epileptic foci for surgical resection, but also to improve understanding of the microstructural changes in long-standing epilepsy. Diffusion tensor imaging (DTI) has the ability to characterize microstructural abnormalities in epileptic foci and to demonstrate the white matter ﬁbers and tracts participating in the epileptic network. DTI is an MRI technique, which is based upon the ability of MRI to assess the direction and magnitude of water diffusion in tissues in vivo by utilizing the principle of anisotropic diffusion of water molecules in the white matter tracts of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with different age groups having temporal lobe epilepsy diagnosed by EEG with no detected structural brain lesion by conventional MRI other than mesial temporal sclerosis.

Exclusion Criteria:

* Contraindications for MRI as claustrophobia, cardiac pacemaker and non-compatible metallic devices.
* Patients with suboptimal images or techniques.
* Post-operative and post-head traumatic cases.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with idiopathic temporal lobe epilepsy and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Hippocampal mean diffusivity (MD) values measured by diffusion tensor imaging (DTI) in patients with temporal lobe epilepsy and non-epileptic control subjects. | Baseline
  Bilateral hippocampal MD values will be measured in square millimeters per second (mm²/s) by diffusion tensor imaging (DTI). MD value of the epileptogenic hippocampus will be compared with the contralateral side and with hippocampal MD values of age- and sex-matched control subjects.

REFERENCES:
- [Background] Caseload survey: CCM certification ranks first. Hosp Case Manag. 2001 Jun;9(6):85-6, 93, 81-2. PMID 11373807
- [Background] Wang Y, Spatz MK, Kannan K, Hayk H, Avivi A, Gorivodsky M, Pines M, Yayon A, Lonai P, Givol D. A mouse model for achondroplasia produced by targeting fibroblast growth factor receptor 3. Proc Natl Acad Sci U S A. 1999 Apr 13;96(8):4455-60. doi: 10.1073/pnas.96.8.4455. PMID 10200283
- [Background] Clark JE, Cant AJ. Lymphadenopathy. Arch Dis Child. 1996 Apr;74(4):368. doi: 10.1136/adc.74.4.368-a. No abstract available. PMID 8669948